CLINICAL TRIAL: NCT06928415
Title: Efficacy and Safety of Liver Transplantation for Hepatocellular Carcinoma With Bile Duct Tumor Thrombus: a Single-arm, Multicenter, Prospective Study (HCC-BDTT in LT)
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT-2024-ZJU-OBS12
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-01

CONDITIONS: Liver Transplant; Hepatocellular Carcinoma; Bile Duct Tumor Thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCC-BDTT in LT: HCC and BDTT patients in LT

SUMMARY:
The prognosis for patients diagnosed with hepatocellular carcinoma with bile duct tumor thrombus (BDTT-HCC) remains notably grim, as there are presently no universally accepted treatment guidelines in place to address this complex condition. Long-term outcomes of liver transplantation (LT) for BDTT-HCC are unclear, whether LT is a proper therapeutic option for BDTT-HCC patients remains to be determined. Therefore, we designed a clinical trial to evaluate survival of BDTT-HCC patients in LT. This is an open-labeled, single-arm, prospective, multicenter and real-world study designed to assess the survival outcomes of BDTT-HCC patients in LT. Patients will be enrolled based on histological confirmation of HCC with BDTT. The study will span a total of 4 years, including a 2-year enrollment phase and a subsequent 2-year follow-up period. We anticipate that LT will provide favorable survival benefits for BDTT-HCC patients, particularly in the key indicator recurrence-free survival (RFS) and improved quality of life. Upon successful completion of the trial, we will extend our monitoring over a longer follow-up time to accurately estimate important indicators such as overall survival (OS). We expect that this study will provide substantial evidence to refine treatment guidelines through thorough data analysis, ultimately contributing to better patient outcomes and advancing our understanding of the disease.

ELIGIBILITY:
Inclusion Criteria:

(1) age between 18 and 70 years; (2) Postoperative pathological diagnosis of HCC with BDTT requiring LT; (3) the general condition can tolerate the operation; (4) written informed consent given by the patient; (5) patients without distant metastasis.

Exclusion Criteria:

(1) Those who did not undergo regular LT for various reasons, split LT, reduced-size LT, simultaneous transplantation, re-transplantation, multiple-organ recipients are excluded; (2) Additional surgical procedures such as pancreaticoduodenectomy were performed; (3) those with other diseases such as active pulmonary tuberculosis, coronary heart disease, renal insufficiency and so on, which affect the therapeutic effect; (4) Extensive abdominal metastasis was found during operation; (5) serious consequences or deaths caused by anesthesia accident during operation; (6) Postoperative death due to other diseases such as traffic accidents, cardiovascular and cerebrovascular accidents; (7) With distant metastasis before operation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC and BDTT patients in LT
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2029-01-10 (Estimated); Study Completion 2029-01-10 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival rate | 2025.1.10-2029.1.10

SECONDARY OUTCOMES:
Overall survival rate | 2025.1.10-2029.1.10

OTHER OUTCOMES:
Tumor recurrence rate | 2025.1.10-2029.1.10